CLINICAL TRIAL: NCT00020072
Title: Gene Expression Analysis in Cutaneous T-Cell Lymphoma
Brief Title: Analysis of Genes Present in Cutaneous T-cell Lymphoma Cells
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Diagnostic
Other Study IDs: CDR0000067694; NCI-00-C-0068; NCT00004546 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2003-03

CONDITIONS: Lymphoma
Keywords: cutaneous T-cell non-Hodgkin lymphoma; mycosis fungoides/Sezary syndrome
MeSH Terms: conditions — Lymphoma; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome

INTERVENTIONS:
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Analyzing genes that are present in cancer cells may be useful in developing better methods to detect, predict, and treat cutaneous T-cell lymphoma.

PURPOSE: Clinical trial to study genes that are present in cutaneous T-cell lymphoma cells.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify gene expression patterns in malignant T cells that can be used to diagnose cutaneous T-cell lymphoma.
* Determine the patterns of gene expression that distinguish normal skin-homing T cells from malignant T cells.

OUTLINE: Patients are stratified by disease (Sezary syndrome vs mycosis fungoides) and prior treatment (yes vs no).

All patients receive a physical examination, and a medical history is taken. Patients with Sezary syndrome undergo leukapheresis. Patients with plaque/tumor stage mycosis fungoides undergo skin biopsy of involved skin. Malignant T cells from blood or skin are then isolated and patterns of gene expression in the malignant T cells are compared to those in normal skin-homing T cells from healthy donors using a "gene chip" (Lymphochip).

Patients are followed annually for 5 years.

PROJECTED ACCRUAL: A total of 40 patients (20 per disease stratum) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven mycosis fungoides with 2 or more plaques or tumors greater than 1 cm in size OR
* Immunologically proven Sezary syndrome with all of the following:

  * Erythroderma
  * Lymphadenopathy
  * T-cell receptor variable beta chain clonality greater than 10% of total lymphocytes by flow cytometry OR
  * CD4+CD7- T-cell fraction that represents greater than 10% of CD4+ T cells

PATIENT CHARACTERISTICS:

Age:

* 18 to 85

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Not pregnant or nursing
* HIV-1 and HTLV-1 negative
* No prior intravenous drug use

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 2 months since prior systemic chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 2 months since prior electron beam radiotherapy

Surgery:

* Not specified

Other:

* At least 2 weeks since prior topical therapy
* At least 2 months since prior photopheresis
* At least 2 months since prior psoralen ultraviolet light (PUVA) or ultraviolet B (UVB) therapy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-03

CONTACTS AND LOCATIONS:
Overall Officials: Sam T. Hwang, MD, PhD, Study Chair — NCI - Dermatology Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States

REFERENCES:
- [Result] Hwang ST, Fitzhugh DJ. Aberrant expression of adhesion molecules by Sezary cells: functional consequences under physiologic shear stress conditions. J Invest Dermatol. 2001 Mar;116(3):466-70. doi: 10.1046/j.1523-1747.2001.01282.x. PMID 11231324